CLINICAL TRIAL: NCT03009786
Title: Cross-cultural and Psychometric Validation Version of the Xerostomia Inventory Into French Language
Brief Title: Validation of the French Version of the Xerostomia Inventory
Acronym: XIvf
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO16109*
Record Dates: First submitted 2016-12-27; First posted 2017-01-04 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Elderly institutionalized subjects or outpatients
  Interventions: Other: Measurement of salivary flow

INTERVENTIONS:
Other: Measurement of salivary flow — A compress of about 0.95 g which is weighed and then placed under the tongue of the subject for 5 minutes. Once the time has elapsed, the compress is weighed, a simple subtraction determines the weight of saliva produced in 5 minutes

SUMMARY:
The main objective of this study is to achieve cross-cultural and psychometric validation of the Xerostomia Inventory initially developed in English language into French Language. This will be achieved in two stages: First, cross-cultural validation, and a second, psychometric validation The cross-cultural validation will be performed according to the methodology of the Institute for Work and Health, according to the recommended six phases. In a second step, the psychometric validation will be done using longitudinal study. Indeed, an observational, longitudinal, and prospective study will be set up. Analysis of the results will help define the feasibility and acceptability of the tool, its validity (content validity, perceived validity, construct validity, concurrent validity, and discriminant validity), its reliability (internal consistency and reproducibility over time). Longitudinal follow-up of patients is expected to also assess the predictive validity and responsiveness.

DETAILED DESCRIPTION:
Medical context:

There is an intra-individual and inter-individual variability in the production of saliva. Various factors influence the production of saliva. Saliva flow tends to decrease with age, sleep, emotional state, and to increase after eating, and during pregnancy. Some drugs increase the salivary flow, others decrease it. Tobacco and alcohol tend to impair the quality of the saliva. Furthermore, 43% of 40-64 years and 61% over 65 take at least one antisialic medication. Lack of saliva can cause problems chewing, swallowing, speaking, and tasting perceptions. There is an increase in the number of oropharyngeal candidiasis that affects feeding behaviors and would be responsible for malnutrition in the elderly, and an increase in the number of caries for subjects still toothed. For edentulous or partially dentate subjects, salivary film plays two roles: the first is to allow adhesion of complete or almost complete dentures; the following is to protect the oral mucosa. In subjects suffering from mouth dryness the denture becomes difficult. In addition, saliva is essential for the first phase of digestion, for the creation of a correct bolus. There are several methods to measure the salivary flow. The most common include:

* The measurement of salivary flow at rest, the subject leaves the saliva in his mouth then allowed to flow slowly and spit into a funnel connected to a graduated tube for either 6 or 12 minutes. This test can be performed either at rest or stimulated using a paraffin cube or citric acid. These tests are long and therefore not suitable for the elderly.
* The salivary flow measurements using a compress weight of about 0.95 g is weighed and then placed under the tongue of the subject for 5 minutes. Once the elapsed time, the pad is weighed, a simple subtraction determines the weight of saliva produced in 5 minutes. This test can be done like the previous one at rest or after stimulation.

Secretion at rest varies authors 0,05mℓ / min 0,4mℓ / min. The mouth dryness is defined by a total salivary flow rate below 0.1 unstimulated +/- 0,1mℓ / min ≤ 0.16 mℓ / min. The salivary potential of hydrogen (pH) varies between 6.5 and 8.5. Decreased salivary flow will cause a decrease in pH and promote the degradation of the oral health status.

Tool: The Xerostomia Inventory is a scale of measurement of xerostomia with eleven items used in daily practice or research, which results in a sum score giving a score representing the severity of the drought oral perceived by the subject. This tool was developed in 1999 and covers both experimental and behavioral aspects of xerostomia, and showed acceptable psychometric characteristics. Today, this tool is available in English, Spanish and Portuguese languages With this study a tool to measure xerostomia will be available in French; it may be used in clinical studies and in the daily practice of the dentist and or speech therapists to obtain a subjective measure of dry mouth, particularly in the elderly who are the most vulnerable subjects consequences of xerostomia. Currently there is no way to measure xerostomia, it is difficult to assess the processes associated with the patient and case treatment administered it is impossible to say whether it is effective or not.

The aim of this study is to achieve cross-cultural and psychometric validation version of the Xerostomia Inventory into French Language.

ELIGIBILITY:
Inclusion Criteria:

* Age: 65 years or more
* Outpatients or nursing home residents
* Speaking French fluently
* Willing to participate to the study

Exclusion Criteria:

* Incapability to understand the instructions or to fill alone the questionnaire
* Under guardianship

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly institutionalized subjects or outpatients aged 65 years or over
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
The psychometric properties of the Xerostomia Inventory measured by questionnaire | month 6
  The Xerostomia Inventory to be validated is an 11-item summated rating scale which combines the responses to 11 individual items into a single continuous scale score which represents the severity of chronic xerostomia; higher scores represent more severe symptoms. Respondents are asked to choose one of five responses: Never: 1 point; Hardly ever: 2 points; Occasionally: 3 points; Fairly often: 4 points; Very often: 5 points; to the following statements referring to the previous 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France